CLINICAL TRIAL: NCT05718063
Title: MAP for Coaches: A Web-Based Musculoskeletal Athletic Injury Prevention Training Course to Increase the Routine Use of Neuromuscular Training Warm-Up Programs
Brief Title: MAP for Coaches: Translating Sports Injury Prevention Knowledge to Youth Sport Coaches
Acronym: MAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Olu Owoeye, PhD, Assistant Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01238
Record Dates: First submitted 2023-01-09; First posted 2023-02-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Dissemination and Implementation; Neuromuscular Training Exercise Warm-up; Technology-Enabled Knowledge Translation
MeSH Terms: conditions — Behavior | interventions — Microtubule-Associated Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full MAP for Coaches eLearning Training Course (Experimental)
  Interventions: Behavioral: MAP for Coaches - Complete Course
- Summarized MAP for Coaches eLearning Training Course (Active Comparator)
  Interventions: Behavioral: Map for Coaches - Overview

INTERVENTIONS:
Behavioral: MAP for Coaches - Complete Course — The MAP for Coaches is an eLearning (web-based) knowledge translation training course aimed at providing youth sport coaches with the evidence-based education and motivation they need to reduce the risk of musculoskeletal injuries in young athletes. Course modules include a description of: (1) musculoskeletal injuries in youth sport; (2) the importance of injury prevention, and instructions on: (1) applying best practices for musculoskeletal athletic injury prevention, including neuromuscular training programs; (2) using behavioral strategies to successfully implement neuromuscular training warm-up programs in coaching sessions.
  Arms: Full MAP for Coaches eLearning Training Course
Behavioral: Map for Coaches - Overview — This is a summarized version of the MAP for Coaches. It comprises a 2-page sport-specific injury prevention e-book (reading) containing an overview of the MAP for Coaches training and an infographic summary.
  Arms: Summarized MAP for Coaches eLearning Training Course

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the MAP for Coaches, a web-based Musculoskeletal Athletic injury Prevention training course, in youth sport coaches. The main question it aims to answer are:

* Is the MAP for Coaches effective in increasing coaches' sport-specific knowledge of musculoskeletal injuries (types, incidence, risk factors, mechanisms, and best prevention practices, with focus on neuromuscular training warm-up exercise programs)?
* Is the MAP for Coaches effective in increasing coaches' motivation (self-efficacy and intention) to use sport-specific neuromuscular training warm-up exercise programs?

The additional questions it aims to answer are:

* Are the effects of the MAP for Coaches sustained in the short- and long-term?
* Is the MAP for Coaches effective in promoting the use of sport-specific neuromuscular training warm-up exercise programs in youth sport coaches?

Regardless of group, participants will receive the MAP for Coaches eLearning training course; however, the participants allocated to the control group will have their post-test survey completed right after they review the sport-specific 2-page injury prevention e-book containing an overview of the MAP for Coaches training course, including an infographic summary (Summarized MAP for Coaches eLearning Training Course). The intervention group will complete the post-test survey after the full training including both the course summary and the detailed course modules (the full training).

The investigators will compare the two groups to see if an exposure to the (Full) MAP for Coaches eLearning Training Course improves study outcomes compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Active and ongoing engagement in team youth sport coaching
* Member of a youth sport organization in the United States
* Must be a team sport coach for one of the following: soccer, basketball, football or volleyball

Exclusion Criteria:

* Additional engagement in adult coaching
* No email address contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge Scores on an 11-Point Likert (0-10) Scale | Baseline, Immediately after online training
  Perceived knowledge regarding sport-specific musculoskeletal injuries and prevention. Minimum value possible is 0 (no knowledge) and maximum value possible is 10 (very high knowledge). Higher scores mean better outcome.
Change in Knowledge Scores Based on 5 Course-Specific Questions (0-5) | Baseline, Immediately after online training
  Objective change in knowledge assessment regarding sport-specific musculoskeletal injuries and prevention based on 5 questions related to the lessons in the training course. Minimum value possible is 0 (poor knowledge score) and maximum value possible is 5 (very high knowledge score). Higher scores mean better outcome.
Change in Self-Efficacy Scores on a 5-Point (1-5) Likert Scale | Baseline, Immediately after online training
  Perceived confidence regarding their ability to implement sport-specific neuromuscular training warm-up exercises. Minimum value possible is 1 (strongly disagree) and maximum value possible is 5 (strongly agree). Higher scores mean better outcome.
Change in Intention Scores on a 5-Point (1-5) Likert Scale | Baseline, Immediately after online training
  Regarding their plan to implement sport-specific neuromuscular training warm-up exercises (self-report). Minimum value possible is 1 (strongly disagree) and maximum value possible is 5 (strongly agree). Higher scores mean better outcome.

SECONDARY OUTCOMES:
Long-term Change in Knowledge Scores on an 11-Point Likert (0-10) Scale | Immediately after online training, 6 months post-training
  Perceived knowledge regarding sport-specific musculoskeletal injuries and prevention. Minimum value possible is 0 (no knowledge) and maximum value possible is 10 (very high knowledge). Higher scores mean better outcome.
Adherence to Neuromuscular Training Warm-up Exercises on a 4-Point (0-3) Likert Scale | 6 months post-training
  Their rate of utilizing sport-specific neuromuscular training warm-up exercises with their team over the past 6 months (self-report). Minimum value possible is 0 (never) and maximum value possible is 3 (always). Higher scores mean better outcome.
Sustained Adherence to Neuromuscular Training Warm-up Exercises on a 4-Point (0-3) Likert Scale | 12 months post-training
  Their rate of utilizing sport-specific neuromuscular training warm-up exercises with their team over the past 12 months (self-report). Minimum value possible is 0 (never) and maximum value possible is 3 (always). Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Olu Owoeye, PhD, Principal Investigator — St. Louis University
Locations (1):
- Olu Owoeye, St Louis, Missouri, United States